CLINICAL TRIAL: NCT03926806
Title: Effect of Dietary Intervention With Dairy Products (Yoghurt) on Body Weight Management and Glycemic Control of T2DM Patients
Brief Title: Yoghurt Consumption, Body Weight Management and Glycemic Control of T2DM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Amalia Yanni, Research and Teaching Associate-Staff, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1354.18-11-16
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: yoghurt; vitamins B; body weight; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain yoghurt (Active Comparator): 2x200g plain yoghurt/day for 12 weeks
  Interventions: Other: Plain yoghurt
- Vitamin B yoghurt (Experimental): 2x200g yoghurt enriched with vitamins B for 12 weeks
  Interventions: Other: Vitamin B yoghurt

INTERVENTIONS:
Other: Plain yoghurt — cups of 200 g yoghurt
  Other Names: Conventional yoghurt
  Arms: Plain yoghurt
Other: Vitamin B yoghurt — cups of 200 g yoghurt
  Arms: Vitamin B yoghurt

SUMMARY:
The study investigates the effects of consumption of yoghurt enriched with vitamins B compared to plain yoghurt, on body weight management and glycemic control of overweight/obese T2DM patients. It also investigates the effect of plain yoghurt consumption on gut hormones response of T2DM patients.

DETAILED DESCRIPTION:
In a large number of epidemiological studies, low-fat dairy consumption has been associated with lower risk of T2DM. However, the number of randomized clinical trials which examine the impact of yoghurt consumption on glycemic control and body weight management of T2DM patients is small and include yoghurts fortified with vitamin D or probiotics. According to our knowledge, fortification of yoghurt with other classes of vitamins beyond vitamin D has not been examined. Vitamins of B-complex hold key-role in energy metabolism. In the state of diabetes mellitus, the requirements for this vitamin class may be higher because of their water solubility and increased excretion. Two groups of patients participated in the study. One group received yoghurt enriched with vitamins B and one group received isocaloric plain yoghurt. In addition, in order to investigate the effect of plain yoghurt on gut hormones, responses to a mixed meal tolerance test were evaluated in the beggining and the end of the dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-36
* HbA1C < 8.5%
* Constant body weight and dietary habits for the last 3 months
* Stable dose of oral medication for at least 3 months
* Diagnosed with T2DM for more than 1 year

Exclusion Criteria:

* History of cardiovascular, gastrointestinal, renal and endocrinological diseases
* Treatment for weight reduction
* Lactose intolerance
* Allergies to milk and dairy products
* Alcohol consumption (> 2 drinks per day)
* Intake of supplements
* Receiving insulin

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Body weight management | 12 weeks
  Change of body weight after dietary intervention
Glycemic control | 12 weeks
  Change of fasting plasma glucose after dietary intervention

SECONDARY OUTCOMES:
Change of ghrelin response | 12 weeks
  Change of ghrelin after the 12 weeks dietary intervention
Change of GLP-1 response | 12 weeks
  Change of GLP-1 after the 12 weeks dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Amalia Yanni, Principal Investigator — Harokopio University; Nikolaos Tentolouris, Study Chair — National and Kapodistrian University of Athens; Vaios Karathanos, Study Director — Harokopio University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panahi S, Tremblay A. The Potential Role of Yogurt in Weight Management and Prevention of Type 2 Diabetes. J Am Coll Nutr. 2016 Nov-Dec;35(8):717-731. doi: 10.1080/07315724.2015.1102103. Epub 2016 Jun 22. PMID 27332081
- [Background] Kaur B, Henry J. Micronutrient status in type 2 diabetes: a review. Adv Food Nutr Res. 2014;71:55-100. doi: 10.1016/B978-0-12-800270-4.00002-X. PMID 24484939
- [Background] El Khoury D, Brown P, Smith G, Berengut S, Panahi S, Kubant R, Anderson GH. Increasing the protein to carbohydrate ratio in yogurts consumed as a snack reduces post-consumption glycemia independent of insulin. Clin Nutr. 2014 Feb;33(1):29-38. doi: 10.1016/j.clnu.2013.03.010. Epub 2013 Mar 27. PMID 23591152